CLINICAL TRIAL: NCT05501249
Title: Effects of Aquatic Integrated Cognitive Motor Training on Cognition and Mobility in Older Adults
Brief Title: Aquatic Exercise for Cognition and Mobility in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emily Dunlap (Other)
Responsible Party: Sponsor-Investigator, Emily Dunlap, Principal Investigator, University of Texas at Austin
Organization: University of Texas at Austin (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00001403
Record Dates: First submitted 2022-08-10; First posted 2022-08-15 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Aging Well; Aging Problems; Cognitive Change; Gait, Unsteady; Mobility Limitation
Keywords: Aquatic exercise; Fall prevention; Functional mobility
MeSH Terms: conditions — Gait Disorders, Neurologic; Mobility Limitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aquatic Exercise Group (Experimental): Aquatic class 45 minutes, 3 times a week, for 8 weeks
  Interventions: Behavioral: Aquatic Integrated Cognitive Motor Training
- Control Group (No Intervention): Usual care for 8 weeks and one hour education session on fall prevention.

INTERVENTIONS:
Behavioral: Aquatic Integrated Cognitive Motor Training — Aquatic exercise class with focus on cognitive and physical exercise
  Arms: Aquatic Exercise Group

SUMMARY:
The purpose of this study is to assess the effects of an aquatic exercise program on cognition and physical function of older adults.

ELIGIBILITY:
Inclusion Criteria:

* Able to ambulate 100 ft independently with or without assistive device
* Score greater than or equal to 3 on the Mini-Cog Test
* Stable medical condition within one month prior to the study
* Stable exercise program within one month prior to the study
* Available during study testing and group class times
* COVID-19 vaccination
* Permission from medical provider to participate in the study

Exclusion Criteria:

* History of dementia or Alzheimer's
* Contraindication to exercise or pool immersion (e.g., unstable cardiovascular conditions, fever, diarrhea, aqua-phobia)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Stroop Effect Test: Change from baseline to the end of intervention/control period | Measures taken at baseline and again at approximately 9-10 weeks
  Measure of working memory and attention
Trail Making Test A and B: Change from baseline to the end of intervention/control period | Measures taken at baseline and again at approximately 9-10 weeks
  Measure of visual scanning and working memory
Digit Backwards Test : Change from baseline to the end of intervention/control period | Measures taken at baseline and again at approximately 9-10 weeks
  Measure of working memory capacity
Gait Measurements: Change from baseline to the end of intervention/control period | Measures taken at baseline and again at approximately 9-10 weeks
  4 gait conditions (single task gait, dual task gait with head turns, dual task gait with head nods, and dual task gait count backwards by serial 7s). Gait measures collected with Strideway Gait Analysis System.
Functional Outcome Measures: Change from baseline to the end of intervention/control period | Measures taken at baseline and again at approximately 9-10 weeks
  Timed Up and Go Test, Cognitive Timed Up and Go Test, Single Leg Balance Test, and Four Square Step Test.

SECONDARY OUTCOMES:
Vital Sign measurements: Change from baseline to the end of intervention/control period | Measures taken at baseline and again at approximately 9-10 weeks
  Blood pressure and heart rate taken after 5 min supine, immediately upon standing, and 2 min after standing
Anthropometric measurements: Change from baseline to the end of intervention/control period | Measures taken at baseline and again at approximately 9-10 weeks
  Height and weight
Neurotrophic Growth Factors: Change from baseline to the end of intervention/control period | Measures taken at baseline and again at approximately 9-10 weeks
  Serum concentration of brain derived neurotrophic factor and insulin-like growth factor 1
Numeric Pain Rating Scale: Change from baseline to the end of intervention/control period | Measures taken at baseline and again at approximately 9-10 weeks
  An 11 point scale for level of pain from 0 (no pain) to 10 (severe pain).
Global Rating of Change Questionnaire: Change from baseline to the end of intervention/control period | Measures taken at baseline and again at approximately 9-10 weeks
  A 15 point global rating scale for changes in domains, from -7 (a great deal worse); through 0 (no change) to +7 (a great deal better).
Activities-specific balance confidence scale: Change from baseline to the end of intervention/control period | Measures taken at baseline and again at approximately 9-10 weeks
  A structured questionnaire that measures an individuals confidence performing daily activities. The minimum score is 0% (no confidence in balance) to 100% (complete confidence in balance).

CONTACTS AND LOCATIONS:
Overall Officials: Emily Dunlap, BS, Principal Investigator — The University of Texas at Austin
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Sharing of deidentified individual participant data will be available upon reasonable request.
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: The data will become available after publication
Access Criteria: Data will be available to researcher for meta-analysis purpose upon reasonable request.

REFERENCES:
- [Background] Carter HH, Spence AL, Pugh CJ, Ainslie P, Naylor LH, Green DJ. Cardiovascular responses to water immersion in humans: impact on cerebral perfusion. Am J Physiol Regul Integr Comp Physiol. 2014 May;306(9):R636-40. doi: 10.1152/ajpregu.00516.2013. Epub 2014 Feb 19. PMID 24553298
- [Background] Bressel E, Louder TJ, Raikes AC, Alphonsa S, Kyvelidou A. Water Immersion Affects Episodic Memory and Postural Control in Healthy Older Adults. J Geriatr Phys Ther. 2019 Oct/Dec;42(4):E1-E6. doi: 10.1519/JPT.0000000000000192. PMID 29738406
- [Background] Parfitt R, Hensman MY, Lucas SJE. Cerebral Blood Flow Responses to Aquatic Treadmill Exercise. Med Sci Sports Exerc. 2017 Jul;49(7):1305-1312. doi: 10.1249/MSS.0000000000001230. PMID 28166116
- [Background] Pugh CJ, Sprung VS, Ono K, Spence AL, Thijssen DH, Carter HH, Green DJ. The effect of water immersion during exercise on cerebral blood flow. Med Sci Sports Exerc. 2015 Feb;47(2):299-306. doi: 10.1249/MSS.0000000000000422. PMID 24977699
- [Background] Kang DW, Bressel E, Kim DY. Effects of aquatic exercise on insulin-like growth factor-1, brain-derived neurotrophic factor, vascular endothelial growth factor, and cognitive function in elderly women. Exp Gerontol. 2020 Apr;132:110842. doi: 10.1016/j.exger.2020.110842. Epub 2020 Jan 15. PMID 31954186
- [Background] Commandeur D, Klimstra MD, MacDonald S, Inouye K, Cox M, Chan D, Hundza SR. Difference scores between single-task and dual-task gait measures are better than clinical measures for detection of fall-risk in community-dwelling older adults. Gait Posture. 2018 Oct;66:155-159. doi: 10.1016/j.gaitpost.2018.08.020. Epub 2018 Aug 23. PMID 30195218
- [Background] de Assis GG, de Almondes KM. Exercise-dependent BDNF as a Modulatory Factor for the Executive Processing of Individuals in Course of Cognitive Decline. A Systematic Review. Front Psychol. 2017 Apr 19;8:584. doi: 10.3389/fpsyg.2017.00584. eCollection 2017. PMID 28469588
- [Background] Doi T, Shimada H, Makizako H, Tsutsumimoto K, Hotta R, Nakakubo S, Suzuki T. Association of insulin-like growth factor-1 with mild cognitive impairment and slow gait speed. Neurobiol Aging. 2015 Feb;36(2):942-7. doi: 10.1016/j.neurobiolaging.2014.10.035. Epub 2014 Nov 1. PMID 25467636
- [Background] Nissim M, Hutzler Y, Goldstein A. A walk on water: comparing the influence of Ai Chi and Tai Chi on fall risk and verbal working memory in ageing people with intellectual disabilities - a randomised controlled trial. J Intellect Disabil Res. 2019 Jun;63(6):603-613. doi: 10.1111/jir.12602. Epub 2019 Feb 18. PMID 30775818
- [Background] Sato D, Seko C, Hashitomi T, Sengoku Y, Nomura T. Differential effects of water-based exercise on the cognitive function in independent elderly adults. Aging Clin Exp Res. 2015 Apr;27(2):149-59. doi: 10.1007/s40520-014-0252-9. Epub 2014 Jun 26. PMID 24965855